CLINICAL TRIAL: NCT00281853
Title: Characterization of Chemotherapy/Biotherapy-Induced Peripheral Neuropathy: Refinement of Clinical Measures
Brief Title: Nerve Changes in Patients Who Are Undergoing Chemotherapy or Biological Therapy for Cancer
Status: Completed | Type: Observational
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Constance Visovsky, PhD, RN, ACNP, Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Other Study IDs: CASE13Z04; P30CA043703 (NIH); CASE-13Z04 (Other: Case Comprehensive Cancer Center); CASE-120411
Record Dates: First submitted 2006-01-24; First posted 2006-01-25 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: Neurotoxicity; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: neurotoxicity; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Neurotoxicity Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: management of therapy complications — Patients undergo a 1-hour peripheral nerve function assessment, including hearing, vibratory sensation, and blood pressure testing, at baseline and then at 4, 8, and 12 weeks during treatment with chemotherapy or biologic therapy.

SUMMARY:
RATIONALE: Learning about the effects of chemotherapy and biological therapy on nerve function may help doctors plan treatment and help patients live more comfortably.

PURPOSE: This clinical trial is studying peripheral neuropathy in patients who are receiving chemotherapy or biological therapy for cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the change in peripheral nerve function in cancer patients during and after treatment with chemotherapy or biologic therapy.
* Determine the clinical measurement of hearing-related air and bone conduction and vibratory sensation in these patients.
* Correlate the changes in orthostatic blood pressure using both the Vasotrac automated blood pressure device and the standard clinical automated blood pressure equipment.
* Determine the patient's perception of hearing quality before and after treatment with chemotherapy or biologic therapy.

OUTLINE: This is a multicenter study.

Patients undergo a 1-hour peripheral nerve function assessment, including hearing, vibratory sensation, and blood pressure testing, at baseline and then at 4, 8, and 12 weeks during treatment with chemotherapy or biologic therapy.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of cancer
* Scheduled to be treated with 1 of the following agents:

  * Cisplatin/paclitaxel combination
  * Biologic therapy with high-dose interferon alfa

PATIENT CHARACTERISTICS:

* Normal vision OR vision corrected with glasses or contact lenses
* No diseases or disorders reducing peripheral nerve function, including any of the following:

  * Diabetes mellitus
  * HIV/AIDS
  * Uremia
  * Spinal injuries
  * Alcoholism
  * CNS problems
* No hearing impairment

PRIOR CONCURRENT THERAPY:

* No prior biologic therapy or neurotoxic chemotherapy

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are receiving chemotherapy or biological therapy for cancer.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2005-03; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Hearing as measured by the Weber test and the Rinne test at baseline, and then weeks 4, 8, and 12 during study treatment | baseline, and then weeks 4, 8, and 12 during study treatment
Vibratory sensation as measured by tuning fork at baseline, and then weeks 4, 8, and 12 during study treatment | baseline, and then weeks 4, 8, and 12 during study treatment
Blood pressure changes at baseline, and then weeks 4, 8, and 12 during study treatment | baseline, and then weeks 4, 8, and 12 during study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Constance Visovsky, PhD, Principal Investigator — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States